# **Hacettepe University Faculty of Medicine**

Department of Anesthesiology and Reanimation

Clinical Trial Study Protocol

Official Title: Comparison of Eleveld and Schnider Target-Controlled Infusion (TCI) Models

for Propofol Sedation in Intensive Care Unit Patients

NCT Number: NCT PENDING

Date: October 28, 2025

Principal Investigator: Assoc. Prof. Başak Akça

Co-Investigators: Prof. Seda Banu Akıncı, Dr. Duygu Özdemir Şimşek

Hacettepe University Hospital, Ankara, Türkiye

## **Background and Rationale**

Evidence-based international guidelines on ICU sedation for mechanically ventilated patients provide similar recommendations. Sedation is routinely administered in critically ill patients to reduce anxiety, facilitate procedures, decrease oxygen consumption and autonomic hyperactivity, and minimize ventilator asynchrony. The goal is to maintain patient comfort and hemodynamic stability while ensuring easy arousability, except in cases requiring deep sedation. Current guidelines recommend using the minimum effective sedation level and performing daily awakening to improve outcomes. Propofol is the preferred sedative due to its rapid onset and predictable recovery. Target-Controlled Infusion (TCI) systems help achieve desired effect-site concentrations based on pharmacokinetic and pharmacodynamic models. The Schnider model is widely used, while the newer Eleveld model integrates broader demographic covariates and has superior predictive performance. This study compares both models in ICU sedation regarding hemodynamic stability, sedation performance, awakening, extubation, ICU discharge, and delirium incidence.

## **Study Objectives**

To compare the clinical performance of the Eleveld and Schnider propofol TCI models in ICU patients regarding hemodynamic stability, sedation performance, awakening and extubation times, delirium incidence, and ICU length of stay.

## **Study Design**

Study Type: Observational (Prospective Cohort Study)

Time Perspective: Prospective

Study Location: Hacettepe University Faculty of Medicine, Department of Anesthesiology

and Reanimation, Intensive Care Unit, Ankara, Türkiye

Study Period: February 2025 – December 2025

Estimated Enrollment: 84 participants (42 per group)

Sampling Method: Consecutive sampling

Two groups will be observed:

- 1. Patients sedated with propofol using the Schnider TCI model.
- 2. Patients sedated with propofol using the Eleveld TCI model.

Sedation with TCI propofol is routine practice in the ICU, and this study will not alter clinical management or drug choice. The responsible anesthesiologist will decide on sedation use independently.

## **Eligibility Criteria**

**Inclusion Criteria:** 

- Age ≥18 years
- ASA I-IV
- Sedation required for mechanical ventilation

- Sedation ≤72 hours
- Informed consent obtained

#### Exclusion Criteria:

- ASA >IV
- BMI ≥35
- Propofol allergy or lipid metabolism disorder
- Sedation >72 hours
- Neurological or neurodegenerative disease affecting consciousness assessment

#### **Outcome Measures**

## Primary Outcome:

- Sedation depth accuracy (BIS 40-60, Riker SAS 3-4)

### **Secondary Outcomes:**

- 1. Hemodynamic stability (MAP, HR)
- 2. Awakening and extubation times
- 3. Delirium incidence (CAM-ICU)
- 4. ICU length of stay
- 5. Adverse events

### **Data Collection and Analysis**

Demographic and clinical data (age, sex, height, weight, comorbidities) will be recorded. Sedation depth will be evaluated every 4 hours using BIS and Riker SAS. Statistical tests: Shapiro–Wilk for normality; Student's t-test or Mann–Whitney U for continuous variables; Chi-square or Fisher's exact test for categorical variables; significance set at p<0.05.

#### **Ethical Considerations**

Approved by the Hacettepe University Clinical Research Ethics Committee. Written informed consent will be obtained. No deviation from standard ICU practice will occur. The study is purely observational.

#### **Research Team**

Principal Investigator: Assoc. Prof. Başak Akça

Co-Investigators: Prof. Seda Banu Akıncı, Dr. Duygu Özdemir Şimşek

Hacettepe University Faculty of Medicine, Department of Anesthesiology and Reanimation.